CLINICAL TRIAL: NCT01824147
Title: ASS-Nonresponse Following Cardiac Surgery as Assessed With Multiple Electrode Aggregometry
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Collaborators: University Hospital Goettingen (Other)
Responsible Party: Principal Investigator, Christian F. Weber, MD, Dr.med. Dr.med. habil Christian F. Weber, Goethe University
Other Study IDs: 33/13
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: ASS-Nonresponse
Keywords: ASS-Nonresponse; cardiac; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG Patients: Patients undergoing surgery for coronary revascularization.

SUMMARY:
It is the aim of the present study to assess the prevalence of ASS-Nonresponse following cardiac surgery using the Multiple Electrode Aggregometry (MEA).

DETAILED DESCRIPTION:
Up to now there are no data concerning the prevalence of ASS-Nonresponse following surgical coronary revascularization procedures as assessed with the Multiple Electrode Aggregometry. Results of the present observational study are needed to assess the prevalence of ASS-Nonresponse in order to perform a sample size analysis for a prospective interventional study in a second step.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years after cardiac surgery
* Antiaggregatory therapy with aspirin postoperatively

Exclusion Criteria:

* known allergy to aspirin
* need for an antiaggregatory therapy other than aspirin
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients following cardiac surgery and a antiaggregatory therapy with aspirin
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ASPItest | at day 3 and 5 after the first dose of aspirin following surgery
  Area under the aggregation curve following stimulation with arachidonic acid in the Multiple Electrode Aggregometry (MEA)

SECONDARY OUTCOMES:
TRAPtest | at day 3 and 5 after the first dose of aspirin following surgery
  Area under the aggregation curve in the Multiple Electrode Aggregometry following stimulation with thrombin receptor activating peptide 6
Platelet Count | at day 3 and 5 after the first dose of aspirin following surgery
  Platelet count taken from the daily standard laboratory results.
Mortality | 12 month
  Mortality will be assessed by a telephonic follow up interview 12 month after enrollment into the study
Myocardial infarction | 12 month
  Occurrence of a myocardial infarction during the 12 month following surgery assessed in a telephonic follow up interview.
Readmission to hospital | 12 month
  Did a readmission to hospital due to cardiac or pulmonary reasons take place in the 12 month following enrollment into the study? Assessed by a telephonic follow up interview.

OTHER OUTCOMES:
Age | at the day of enrollment
  Age of the patient in years at the time of enrollment
Height | at the day of enrollment
  Height of the patient in centimeters at the time of enrollment
Weight | at the day of enrollment
  Weight of the patient in kilograms at enrollment
Gender | at the day of enrollment
  Gender of the patient
LDL cholesterol | at the day of enrollment
  LDL cholesterol of the patient in mg/dl at enrollment
nicotine | at the day of enrollment
  Smoking habits of the patient will be documented at enrollment in the categories:
  * active smoker
  * non smoker
European system for cardiac operative risk evaluation (EuroSCORE) | at the day of enrollment
  EuroSCORE as assessed on admission will be documented.
Diabetes | at the day of enrollment
  Risk factor diabetes will be documented in the following categories at enrollment:
  * Diabetes Typ I
  * Diabetes Typ II without the need for insulin substitution
  * Diabetes Typ II with the need for insulin substitution
Surgical procedure | at the day of enrollment
  The surgical procedure performed will be documented.
phone number | at the day of enrollment
  The phone will be documented for the 12 month follow up interview.

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, MD, Principal Investigator — Goethe University Frankfurt
Locations (2):
- Germany (2):
  - Goethe - University, Frankfurt am Main, Hesse
  - University Hospital Goettingen, Göttingen, Lower Saxony

REFERENCES:
- [Background] Collet JP, Cuisset T, Range G, Cayla G, Elhadad S, Pouillot C, Henry P, Motreff P, Carrie D, Boueri Z, Belle L, Van Belle E, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Barthelemy O, Beygui F, Silvain J, Vicaut E, Montalescot G; ARCTIC Investigators. Bedside monitoring to adjust antiplatelet therapy for coronary stenting. N Engl J Med. 2012 Nov 29;367(22):2100-9. doi: 10.1056/NEJMoa1209979. Epub 2012 Nov 4. PMID 23121439